CLINICAL TRIAL: NCT04747002
Title: Investigator-initiated Clinical Trial (Phase II) of Cancer Vaccine "DSP-7888" for Acute Myeloid Leukemia Patients.
Brief Title: Investigator-initiated Clinical Trial (Phase II) of Cancer Vaccine "Dainippon Sumitomo Phama(DSP)-7888" for Acute Myeloid Leukemia Patients.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Yoichi Yamamoto, Professor, Osaka University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WT1-AM-05
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia in Remission

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration Group (Active Comparator): Patients who are injected with DSP-7888.
  Interventions: Drug: DSP-7888
- Non-administration Group (No Intervention): Patients who are only under observation.

INTERVENTIONS:
Drug: DSP-7888 — Cocktail peptide vaccine designed to induce cytotoxic T lymphocytes that recognize WT1 peptides
  Arms: Administration Group

SUMMARY:
This study is an investigator-initiated clinical trial (Phase II) using DSP-7888 for acute myeloid leukemia patients with 1st hematological complete remission (CR). DSP-7888 is a novel cocktail peptide vaccine designed to induce cytotoxic T lymphocytes that recognize Wilms Tumor Gene 1 (WT1) peptides.

DETAILED DESCRIPTION:
This study is an investigator-initiated clinical trial (Phase II) using DSP-7888 for acute myeloid leukemia patients with 1st hematological CR. DSP-7888 is a novel cocktail peptide vaccine designed to induce cytotoxic T lymphocytes that recognize WT1 peptides. Primary endpoint is relapse-free survival, and 2nd endpoint is hematological relapse-free survival, overall survival and adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. acute myeloid leukemia defined by World Health Organization (WHO) 2016 classification
2. favorable or intermediate risk based on European Leukemia Net (ELN) 2017 risk classification
3. 1st hematological after chemotherapy
4. Human Leukocyte Antigen (HLA)-A*02:01, 02:06, 24:02
5. 20-80 years old
6. Eastern Cooperative Oncology Group (ECOG) performance Status 0-2
7. within 35 days after White Blood Cell (WBC) and Neutrophil recovers over 1500 and 500, respectively
8. sufficient organ function as below within 7 days

(1) Neutrophil : >= 1000 (2) Cr : >= 3.0mg/dl (3) Aspartate aminotransferase (AST), Alanine transaminase (ALT) : 5 x the upper limit of normal (ULN) for the reference lab (4) Percutaneous oxygen saturation (SpO2): >= 95% 9) patients who agree contraception until 6 months after the last injection 10) non-candidate for hematopoietic stem cell transplantation.

1. illegible for hematopoietic stem cell transplantation (HSCT)
2. lack of appropriate donor
3. patients who don't select HSCT at the 1st hematological complete remission (hCR) timing

Exclusion Criteria:

1. multiple primary cancer
2. autoimmune disease
3. usage of investigational or unapproved drug within 28 days
4. severe organ failure
5. Human Immunodeficiency Virus (HIV) antibody / Hepatitis B surface (HBs) antigen / Hepatitis C Virus (HCV) antibody positive
6. pregnant woman
7. lactating woman
8. under treatment against active infection
9. difficult to enroll because of mental problem
10. other reasons which investigator judge appropriate for enrollment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | 2 year

SECONDARY OUTCOMES:
Hematological relapse-free survival | 2 year
Overall survival | 2 year
Adverse event | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka University, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://sahswww.med.osaka-u.ac.jp/~hmtonc/vaccine/AM05.html